CLINICAL TRIAL: NCT04360109
Title: Study of the Association Between Presbycusis With the Incidence of Frailty. Intake of Polyphenols for the Prevention of Presbycusis: Effects on Frailty
Brief Title: Study of the Association Between Presbycusis With the Incidence of Frailty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Carolina Sánchez Rodríguez, Principal Investigator, Universidad Europea de Madrid
Other Study IDs: PI19/01524
Record Dates: First submitted 2020-03-09; First posted 2020-04-24 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Presbycusis; Frailty Syndrome; Oxidative Stress
MeSH Terms: conditions — Presbycusis; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the project is to establish the association between presbycusis and the incidence of frailty in humans in order to establish hearing loss with age as another index for the diagnosis of frailty; As well as studying the effect of exposure to polyphenols in the diet on presbycusis and frailty. Human study: volunteers between 60 and 99 years old, men and women during a period of 6 months, questions and answers, audiometries, study of fragility, analysis of antioxidants in blood, and samples of urine will be measured Total polyphenols and oxidant capacity.

ELIGIBILITY:
Inclusion Criteria:

* Age

Exclusion Criteria:

* Disease of the hearing system
* Serious illness (e.g. tumor)
* Dementia
* Total dependence

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who meet the inclusion and exclusion criteria and who attend the ENT or geriatrics clinic
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Auditory function | 6 months
  study by pure tone audiometry, calculating an average of the thresholds of hearing at 0.5, 1, 2 and 4 kilohertz classifying according to their hearing thresholds to the participants in: normal hearing ≤ 25decibel, slight hearing loss = 26-40 decibel; Y moderate-greater hearing loss> 40 decibel (according to the World Health Organization).
Frailty | 6 months
  Fragility will be determined at the beginning and at the end of the study period using the 5 Fried indexes: weakness, low speed, low physical activity, exhaustion and weight loss. Participants with 3 or more criteria are classified as fragile, with 1-2 criteria as pre-fragile, and those without any criteria are not considered fragile.
  Thus, individuals will be classified in the analyzes as non-fragile, pre-fragile and fragile.

SECONDARY OUTCOMES:
Determination of total polyphenols in urine | measured twice in each volunteer, at the beginning and end of the study period (6 months)
  24-hour urine samples using the method Folin -Ciocalteu.
Blood analysis, | It will be performed at the beginning and at end of the study period (6 months)
  routine biochemistry and determination of: carotenoids, vitamins E and D
Microbiota | It will be performed at the beginning and at end of the study period (6 months)
  Stool microbiota analysis

CONTACTS AND LOCATIONS:
Overall Officials: Carolina S Rodríguez, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Hospital Universitario de Getafe, Getafe, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided